CLINICAL TRIAL: NCT00351065
Title: an 8week, Multi-Center, Randomized, Double Blind, Placebo-Controlled,Parallel Group, Fixed Dose, Dose-Finding Study to Assess the Efficacy and Safety of SK3530 in Patients With Erectile Dysfunction.
Brief Title: Phase II Trial of SK3530 in Erectile Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK3530_II_2004
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-07

CONDITIONS: Male Erectile Dysfunction
Keywords: erectile dysfunction, PDE-5 inhibitor
MeSH Terms: conditions — Erectile Dysfunction | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride

INTERVENTIONS:
Drug: SK3530

SUMMARY:
This study was designed to evaluate the efficacy and safety of the SK3530 tablet and to find the optimal dose and dosage schedule after oral administration to patients with erectile dysfunction.

DETAILED DESCRIPTION:
Double-blind, Placebo-controlled, randomized, parallel group, fixed dose, multi-center dose-finding study.

The patients voluntarily signed the informed consent form of the clinical study and underwent a screening. After completing the four-week run-in period, they were randomly assigned to either a placebo group or one of the three SK3530 groups: 50mg, 100mg, and 150mg. The study was conducted in a double-blind manner. A different dose of SK3530 was administered to the subjects depending on the assigned treatment group for 8 weeks. Patient's visit took place at week 4 and week 8 after randomization and at 6 or 7days after end of study.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 19 to 70, suffering from erectile dysfunction for at least the past six months.

Definition of erectile dysfunction: "the inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance."

* Subjects who had a stable, heterosexual relationship with a single partner.
* In the case of the sex partner being of childbearing potential age, the partner having consented to use a medically reliable contraceptive such as the pill, injection, or intrauterine device throughout the whole study period. Not applicable if the sex partner was surgically sterilized, underwent hysterectomy, or was one of the cases that were assessed as acceptable by an investigator.
* Subjects who are eligible for study subjects in the screening test.
* Subjects who attempted sexual intercourse four times or more but failed at least 50% of the attempts or more during the four-week run-in period
* Subjects who had 5~22 scores in the IIEF EF domain during the four-week run-in period
* Subjects who voluntarily decided to participate in the study and sign the informed consent form

Exclusion Criteria:

* Subjects who had spinal injury or radical prostatectomy
* Subjects who has anatomical deformities of penis (e.g. severe penile fibrosis, Peyronie's disease)
* Subjects who are diagnosed as primary hypoactive sexual desire
* Erectile dysfunction due to neurogenic or endocrine disorders such as hyperprolactinemia, low testosterone, etc.

Hyperprolactinemia: blood prolactin level ≥ 3 X upper limit of normal Low testosterone: blood total testosterone level < lower limit of normal

* Subjects who has major psychiatric disorder (including major depression or schizophrenia), and significant neurology disorders (such as neurovascular disorder, etc.) that is not well controlled on treatment
* Known history of alcoholism or substance abuse.
* Hepatic and renal disease Hepatic disease: GOT, GPT ≥ 3 X upper limit of normal Renal disease: blood creatinine ≥ 2.5mg/dl
* Currently uncontrolled diabetes mellitus (HbA1C>12%)
* Untreated proliferative diabetic retinopathy
* History of stroke, transient ischemic attacks, myocardial infarction, unstable angina, life-threatening arrhythmia, or coronary artery bypass graft surgery within the previous six months
* History of Heart failure of NYHA Class III or IV, or NYHA Class II within the previous six months.
* Hypotension (a resting sitting blood pressure <90/50 mmHg) or uncontrolled malignant hypertension (a resting sitting blood pressure >170/100mmHg)
* A blood disease that might cause a priapism, such as sickle cell disease, multiple myeloma, or leukemia
* Known history of retinitis pigmentosa
* History of serious intestinal bleeding disorder within the past year
* Subjects who had been prescribed Viagra®, Cialis®, Levitra®, intracavernosal injection or other medication to treat erectile dysfunction within the one week prior to screening.
* Subjects who are taking one of the following:

  * Nitrates/Nitric oxide (NO) donors (e.g. nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, amyl nitrate/nitrite, sodium nitroprusside)

    * Anticoagulant (except for anti-platelet agent)

      * Medicines affecting on CYP3A4 metabolism (e.g. erythromycin, itraconazole, ketoconazole, ritonavir, saquinavir, amprenavir, indinavir, nelfinavir, cimetidine)

        * Androgens (e.g. testosterone) or Anti-androgens

          * Trazodone
* Known allergic hypersensitivity to other PDE-5 inhibitors such as Viagra®, Cialis®, Levitra®
* Known no responder to previous treatment with Viagra®, Cialis® or Levitra®
* Subjects who had taken other clinical trial medicine (including a placebo treatment) within the previous 30 days.
* Subjects who are unable or unwilling to keep a patient diary
* Subjects who illiterate or unable to understand questionnaires or a patient diary
* Subjects who have any other clinical condition, which would interfere with the assessment of study results, in the opinion of the investigator

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-09; Study Completion 2005-03

PRIMARY OUTCOMES:
IIEF Q3 & Q4

SECONDARY OUTCOMES:
① Other IFF Questions: Assessment by Domain
② SEP Q2 & Q3: Based on the patient's diary
* SEP: Sexual Encounter Profile
③ GEAQ(Global Efficacy Assessment Question)
: Did the last 4-week treatment improve your erectile function?

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Seung Paick, Doctor, Principal Investigator — Seoul National Univ. Hospital